CLINICAL TRIAL: NCT03638518
Title: Effectiveness of Acupuncture vs. Core Stability Based Physiotherapy in Balance and Functional Capacity of Women With Fibromyalgia: A Randomized Controlled Trial
Brief Title: Acupuncture vs. Core Stability Training in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, Profesor of Physiotherapy, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79/2013
Record Dates: First submitted 2018-08-14; First posted 2018-08-20 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Fibromyalgia
Keywords: rehabilitation; balance; functional capacity; quality of life; pain; acupuncture
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Participants were randomized to a core stability training physiotherapy programme group, an acupuncture treatment group and control group for a 13 week study.
Who Masked: Outcomes Assessor
Masking Description: Neither the participants nor their therapists were blind to the treatment allocation. However, the assessor was independent to the study and was not aware of the treatments applied or the objective of the therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): In the acupuncture experimental group, the technique applied included the use of the following acupuncture points of Traditional Chinesse Medicine: GV20, ST36 and BL60 . One needle insertion was performed in each session and in the case of the last two points the needle insertions were done bilaterally.
  Patients laid supine on a treatment table with their legs exposed. The skin on the acupuncture points was prepared with 70% ethyl alcohol. One-time-use disposable sterile stainless steel needles (0,26x50mm) were inserted into acupuncture points.
  After insertion, acupuncture needles were manually manipulated to obtain the de qi sensation. The needles remained in place for 20 minutes and there were no further manipulations during the retention time.
  Interventions: Other: Acupuncture
- Physiotherapy (Experimental): The physiotherapy experimental group received core stability based physiotherapy treatment. Before the beginning of the treatment sessions, the basic principles of core stability exercises were explained to the participants. The exercise programme included 7 exercises. The exercises in the crook lying position were core activation with breathing, single leg lift with knees bent, single leg slides, bridging and knee drop sideways. The exercises completed in side lying included hip external rotation with knees bent and hip abduction with knees straight. After each session gentle stretching of the lower limbs and lumbar spine were performed. The sessions were administered twice a week during 30 minutes with groups of no more than 8 people.
  Interventions: Other: Physiotherapy
- control (No Intervention): The control group did not receive any intervention. The participants continued with their routine medical treatment.

INTERVENTIONS:
Other: Acupuncture — Acupuncture 5 weeks treatment. 2 sessions a week (30 minutes each session)
  Arms: Acupuncture
Other: Physiotherapy — Core stability exercises programme. 2 sessions a week (30 minutes each session) during 5 weeks
  Arms: Physiotherapy

SUMMARY:
This study analyse the effectiveness of a core stability training Physiotherapy programme versus Acupuncture treatment for the management of balance and functional capacity impairments of women with Fibromyalgia.

DETAILED DESCRIPTION:
Objective:

This study investigated the effectiveness of a core stability training Physiotherapy programme versus Acupuncture for the management of balance and functional capacity impairments of women with Fibromyalgia.

Design:

A single-blind randomized clinical controlled trial.

Setting:

University of Extremadura and Olivenza Fibromyalgia Association, Spain

Subjects:

Women with Fibromyalgia and balance impairment.

Interventions:

135 Participants were randomized to a core stability training physiotherapy programme group (n=45), an acupuncture treatment group (n=45) and control group (n=45) for 13 weeks.

Main Measures:

Measures were taken at baseline (week 0), post intervention (week 6) and at follow up (week 13). The primary outcome measures were static balance (posturography) and dynamic balance and functional mobility (Berg Balance Test, Time Up and Go test and 10-metre walk) and functional capacity (Fibromyalgia Health Assessment Questionnaire (FHAQ) and the physical function item from the Spanish Fibromyalgia Impact Questionnaire (SFIQ)).The secondary outcome measure were quality of life (Spanish- Fibromyalgia Impact Questionnaire), pain, joint stiffness, difficulty to work and depression (measured with the visual analogue scale).

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 71 years old,
* diagnosed with Fibromialgia by a specialized physician,
* having subjective sensation of balance impairments.

Exclusion Criteria:

* The exclusion criteria were to present any medical contraindication for acupuncture and/or physiotherapy, phobia of needles, adverse reactions to medication that could influence in balance, associated pathologies such as alcoholism or severe visual deficit, to have receive acupuncture or core stability based physiotherapy in the two months previous to the intervention and to do physical exercises that train core stability such as Pilates or Yoga

Ages: 18 Years to 71 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — One of the inclusion criteria was to be a woman
Enrollment: 160 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Change from the centre of gravity at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  Static balance and postural control is the ability to maintain the centre of gravity within the base of support. Centre of gravity is measured in percentage through posturography study
Change from the monopodal stance test at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  Static balance and postural control is the ability to maintain the centre of gravity within the base of support. Monopodal stance test measures static balance in percentage through posturography study.
Change from Berg Balance Scale at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  Dynamic balance is the ability to maintain the centre of gravity within the base of support during the performance of functional activities. Berg Balance scale measures dynamic balance through performing multiple tasks and with a score of 0 to 56.
Change from Time Up and Go test at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  Time up and Go test measures dynamic balance showed in seconds
Change from 10 meter walk test at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  10 meter walk test measures walking speed and performance which is related to dynamic balance. The unit use is meter/second.
Change from Health Assessement Questionnaire at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  Health Assessement questionnaire measures the functional capacity of a subject. It provides an impairment score of 0 to 3.
Change from physical function item of the Spanish Fibromyalgia Impact Questionnaire at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The physical function item of the Spanish Fibromyalgia Impact Questionnaire measures functional capacity with a score of 0 to 3.

SECONDARY OUTCOMES:
Change from the Spanish Fibromyalgia Impact Questionnaire at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The Spanish Fibromyalgia Impact Questionnaire measures the quality of life and the impact of Fibromyalgia on the life of persons diagnosed with this condition. The maximum score is 100 and the higher the result obtained, the higher the impact of the condition on the person and the less quality of life he/she has.
Change from pain intensity levels measured with the visual analogue scale at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The visual analogue scale is a 100-mm scale, where 0 indicated 'no symptoms' and 100 indicating 'extreme and unbearable symptoms'.
Change from joint stiffness levels measured with the visual analogue scale at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The visual analogue scale is a 100-mm scale, where 0 indicated 'no symptoms' and 100 indicating 'extreme and unbearable symptoms'.
Change from depression level measured with the visual analogue scale at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The visual analogue scale is a 100-mm scale, where 0 indicated 'no symptoms' and 100 indicating 'extreme and unbearable symptoms'.
Change from perceived difficulty to work measured with the visual analogue scale at 5 weeks and 13 weeks | Before treatment, after 5 weeks of treatment and after 6 weeks of follow up
  The visual analogue scale is a 100-mm scale, where 0 indicated 'no difficulty' and 100 indicating 'extreme and unbearable difficulty'.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mª Garrido Ardila, Professor, Principal Investigator — University of Extremadura

IPD SHARING:
Plan to Share IPD: No